CLINICAL TRIAL: NCT03124212
Title: Cascade Genetic Testing for Hereditary Breast/Ovarian Cancer and Lynch Syndrome in Switzerland
Acronym: CASCADE
Status: Recruiting | Type: Observational
Sponsor: University of Basel (Other)
Collaborators: Kantonal Spital Solothurn, Olten (Unknown); Kantonal Spital Wallis, Sion (Unknown); Kantonal Hospital Lucerne (Unknown)
Responsible Party: Principal Investigator, Maria Katapodi, Professor of Nursing Science, University of Basel
Other Study IDs: 2016-02052
Record Dates: First submitted 2017-04-10; First posted 2017-04-21 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Breast and Ovarian Cancer; Lynch Syndrome
Keywords: mutation carrier; blood relative; genetic testing; family-based cohort
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: CASCADE genetic screening — Family-based cohort of mutation carriers, blood relatives who test negative, and untested blood relatives

SUMMARY:
Breast, colorectal, ovarian, and endometrial cancers constitute approximately 30% of newly diagnosed cancer cases in Switzerland and affect more than 12,000 individuals annually. Several hundred of these patients are likely to carry known genetic mutations associated with HBOC or LS. Genetic testing for hereditary susceptibility to cancer can prevent many cancer deaths through early identification and engagement in high-risk management care that involves intensive surveillance, chemoprevention and/or prophylactic surgery. However, current rates of genetic testing indicate that many Swiss mutation carriers and their family members do not use cancer genetic services (counseling and/or testing), either due to lack of coordination of care or due to lack of communication about the mutation among family members.

Cascade screening identifies and tests family members of a known mutation carrier. It determines whether asymptomatic family members are carriers of the identified mutation and proposes management options to reduce harmful outcomes. Robust evidence of basic science and descriptive population-based studies in Switzerland support the necessity of cascade screening for HBOC and LS. However, translation of this knowledge into public health interventions is lacking.

Specific Aims of the CASCADE study are:

1. Survey Index Patients diagnosed with HBOC or LS from clinic-based genetic testing records and determine their cancer status and surveillance practices; needs for coordination of medical care; psychosocial needs; patient-provider and patient-family communication needs; quality of life; willingness to serve as advocates for cancer genetic services for blood relatives.
2. Survey first- and second-degree relatives, and first cousins identified from pedigrees and/or family history records of HBOC and LS Index Patients and determine their cancer and mutation status; cancer surveillance practices; needs for coordination of medical care; barriers and facilitators to using cancer genetic services; psychosocial needs; patient-provider and patient-family communication needs; quality of life; willingness to participate in a study designed to increase use of cancer genetic services.
3. Explore the influence of patient-provider communication about genetic cancer risk on patient-family communication and the acceptability of a family-based communication, coping, and decision support intervention with focus group(s) of mutation carriers and blood relatives.

DETAILED DESCRIPTION:
Please see study protocol provided in the references

ELIGIBILITY:
Inclusion Criteria:

1. Carrier of a mutation associated with HBOC or LS
2. Have at least one living blood relative
3. Men and women
4. 18 years old and older
5. Mentally and physically able to provide informed consent
6. Can read and speak German or French or Italian or English
7. Currently living in Switzerland.

Exclusion Criteria:

1. Carriers of unclassified variants (VUS) in BRCA1, BRCA2 or MLH1, MSH2, MSH6, PMS2, EPCAM genes
2. Not living in Switzerland
3. Patients who are critically ill and cannot complete the CASCADE survey
4. Participants who are institutionalized (e.g., nursing homes) or incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living carriers of pathogenic mutations associated with HBOC and LS, and their blood relatives (first- and second-degree, and first cousins)
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Establishing the CASCADE Cohort | 12 months
  Response rate for Index Patients with HBOC and LS and blood relatives

SECONDARY OUTCOMES:
Cancer Surveillance | 12 months
  Number of mammograms, CBEs and MRIs of Index Patients and Blood Relatives

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Katapodi, PhD, Principal Investigator — University of Basel
Locations (9):
- Switzerland (9):
  - HFR Fribourg - Hôpital Cantonal, Fribourg, Canton of Fribourg
  - Hirslanden Clinic Des Grangettes, Geneva, Canton of Geneva
  - Hôpital du Jura Service d'Oncologie, Delémont, Canton of Jura
  - Katonsspital Winterthur Tumorzentrum Brustzentrum, Winterthur, Canton of Zurich
  - University Hospital Basel, Basel
  - Istituto Oncologico della Zvizzera Italiana, Bellinzona
  - Gastroenterology clinic, Bern
  - Universitatklinik fur Medizinische Onkologie, Inselspital, Bern
  - Unite d'Oncogenetique et de Prevention des Cancers, Geneva

IPD SHARING:
Plan to Share IPD: Yes
Upon request, including purpose and expected timeline, anonymized patient data will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2024- December 2029
Access Criteria: Upon request - TBD

REFERENCES:
- [Background] Katapodi MC, Viassolo V, Caiata-Zufferey M, Nikolaidis C, Buhrer-Landolt R, Buerki N, Graffeo R, Horvath HC, Kurzeder C, Rabaglio M, Scharfe M, Urech C, Erlanger TE, Probst-Hensch N, Heinimann K, Heinzelmann-Schwarz V, Pagani O, Chappuis PO. Cancer Predisposition Cascade Screening for Hereditary Breast/Ovarian Cancer and Lynch Syndromes in Switzerland: Study Protocol. JMIR Res Protoc. 2017 Sep 20;6(9):e184. doi: 10.2196/resprot.8138. PMID 28931501
- [Background] Nikolaidis C, Ming C, Pedrazzani C, van der Horst T, Kaiser-Grolimund A, Ademi Z, Buhrer-Landolt R, Burki N, Caiata-Zufferey M, Champion V, Chappuis PO, Kohler C, Erlanger TE, Graffeo R, Hampel H, Heinimann K, Heinzelmann-Schwarz V, Kurzeder C, Monnerat C, Northouse LL, Pagani O, Probst-Hensch N, Rabaglio M, Schoenau E, Sijbrands EJG, Taborelli M, Urech C, Viassolo V, Wieser S, Katapodi MC; for the CASCADE Consortium. Challenges and Opportunities for Cancer Predisposition Cascade Screening for Hereditary Breast and Ovarian Cancer and Lynch Syndrome in Switzerland: Findings from an International Workshop. Public Health Genomics. 2018;21(3-4):121-132. doi: 10.1159/000496495. Epub 2019 Jan 29. PMID 30695780
- See also: CASCADE website — https://swisscascade.ch/en/